CLINICAL TRIAL: NCT02058901
Title: A Phase I Study of High-dose, Intermittent Sunitinib in Patients With Solid Tumors.
Brief Title: Study of High-dose, Intermittent Sunitinib in Patients With Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.M.W. Verheul, Prof. Dr., Amsterdam UMC, location VUmc
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2013/75; 2012-005756-41 (EudraCT Number)
Record Dates: First submitted 2013-09-30; First posted 2014-02-10 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Solid Tumors
Keywords: sunitinib; solid tumors
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sunitinib high dose, weekly schedule (Experimental): Initial dose of sunitinib is set at 200 mg once weekly. Three patients are treated at the current dose level. If at least 2 patients are observed to have Dose Limiting Toxicity (DLT), the prior dose level is defined as the Maximum Tolerated Dose (MTD) (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 patients are observed to have DLT, the dose level is escalated one step for the next cohort of 3 patients. If exactly 1 of the 3 patients treated show DLT, 3 additional patients are treated at the current dose level. If none of these show DLT, the dose level is escalated for the next cohort of 3 patients; otherwise, the prior dose level is defined as the MTD (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). A tentative MTD becomes final when a total of 6 patients are treated with less than 2 showing DLT
  Interventions: Drug: Sunitinib
- Sunitinib high dose, biweekly schedule (Experimental): When the final MTD is reached for the cohort of patients treated once weekly and depending on the toxicities developed and defining MTD, enrollment of patients in the once every 2 weeks escalation cohort will begin, with the initial dose set at the MTD dose of the once weekly schedule, escalating again at 100 mg increments per dose level.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib

SUMMARY:
The primary objective of this study is:

* To determine the maximum tolerated dose (MTD) of sunitinib when administered once weekly or once every two weeks.
* To assess the safety and tolerability of sunitinib in a once weekly or once every two weeks dose schedule.

DETAILED DESCRIPTION:
Our hypothesis is that sunitinib, when given in a high-dose, intermittent schedule may exhibit improved efficacy with an acceptable toxicity profile. In the present phase I trial, we aim to determine the maximum tolerated dose of sunitinib when administered high-dose, once weekly or once every two weeks. Furthermore, by acquiring skin and tumor biopsies, we will assess intratumoral concentrations of sunitinib, correlate these to skin and plasma concentrations and gain more insight into the biological effects of the drug. Additionally, we aim to preliminary assess the efficacy of sunitinib administered at the MTD level in both schedules. Known serum angiogenesis markers will be correlated to efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Signed (by the patient or legally acceptable representative) and dated Informed Consent Form
* Histological or cytological documentation of incurable locally advanced or metastatic solid malignancy for which no standard therapy exists.
* Primary tumor or metastatic site must be accessible for biopsy. Patients eligible for the expansion cohort must be willing to undergo tumor biopsies, while tumor biopsy remains optional for patients enrolled in the escalation cohort. Bone metastases are excluded as a biopsy site.
* Evaluable disease by RECIST version 1.1 criteria (see appendix III; at least 1 target or non-target lesion for dose escalation cohorts; at least 1 target lesion for dose expansion cohort).
* Patients must have documented radiographic or clinical progressive disease.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Normal 12-lead ECG (clinically insignificant abnormalities permitted), and Left Ventricular Ejection Fraction (LVEF) > 50% by multigated acquisition (MUGA) scan or echocardiogram.
* Normal regulated thyroid function- suppletion or blocking drugs permitted.
* Urinalysis: no clinically significant abnormalities.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 14 days prior to screening:

  1. Hemoglobin >= 5.6 mmol/l
  2. Absolute neutrophil count (ANC) >=1,5 x 10*9/l
  3. Platelet count >= 100 x 10*9/l
  4. Total bilirubin <=1.5 times the upper limit of normal (ULN)
  5. ALT and AST 2.5 x ULN (In case of liver metastases: < 5 x ULN)
  6. Alkaline phosphatase < 4 x ULN
  7. Serum creatinine <= 1.5 x ULN or Creatinine clearance >= 50 ml/min (based on MDRD)
  8. PT-INR/PTT < 1.5 x ULN, unless coumarin derivatives are used
  9. Activated partial thromboplastin time < 1.25 x ULN (therapeutic anticoagulation therapy is allowed, if this treatment can be interrupted for a biopsy as judged by the treating physician)
* Patients with known Gilbert's disease who have serum bilirubin <= 3x ULN may be enrolled.
* Pregnant or breast-feeding subjects: Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. For fertile men or women of childbearing potential: documented willingness to use a highly effective means of contraception (e.g., hormonal methods [implants, injectables, or combined oral contraceptives], intrauterine devices, sexual abstinence, or vasectomized or surgically sterilized partner). Contraception is necessary for at least 6 months after receiving the study kinase inhibitor.

Exclusion Criteria:

* Evidence of a significant uncontrolled concomitant disease, such as cardiovascular disease (including stroke, New York Heart Association Class III or IV cardiac disease or myocardial infarction within 6 months prior to screening, unstable arrhythmia, clinically significant valvular heart disease and unstable angina); nervous system, pulmonary (including obstructive pulmonary disease and history of symptomatic bronchospasm), renal, hepatic, endocrine, or gastrointestinal disorders; or a serious non-healing wound or fracture.
* Poorly controlled hypertension despite adequate blood pressure medication. Blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen. Blood pressure must be stable on at least 2 separate measurements.
* Seizure disorders requiring anticonvulsant therapy.
* jor surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery.
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including HIV and atypical mycobacterial disease, but excluding fungal infection of the nail beds.)
* Known hypersensitivity to sunitinib or to its excipients.
* Presence of any significant central nervous system or psychiatric disorder(s) that would interfere with the patient's compliance.
* Drug or alcohol abuse.
* Females who are pregnant or breast-feeding.
* Any evidence of a disease or condition that might affect compliance with the protocol or interpretation of the study results or render the patient at high risk from treatment complications.
* Unwillingness or inability to comply with study and follow-up procedures.
* No chemotherapy, radiotherapy, or biologic therapy within the previous 4 weeks; no nitrosoureas or mitomycin C within the previous 6 weeks; no investigational agents within the previous 4 weeks.
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
* Untreated or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control);
* Patients with a history of treated CNS metastases are eligible, provided that all of the following criteria are met:

  1. Presence of evaluable or measurable disease outside the CNS
  2. Radiographic demonstration of improvement upon completion of CNS-directed therapy and no evidence of interim progression between completion of CNS-directed therapy and the screening radiographic study
  3. Completion of radiotherapy ≥ 8 weeks prior to the screening radiographic study
  4. Discontinuation of corticosteroids and anticonvulsants ≥ 4 weeks prior to the screening radiographic study.

Note: Prior sunitinib therapy does not constitute an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-07; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) of sunitinib | 6 weeks
Number of participants with serious and non-serious adverse events | 6 weeks

SECONDARY OUTCOMES:
Calculation of maximum plasma drug concentration, sunitinib half life, Area Under the Concentration-Time Curve (AUC 0-48h), clearance and volume of distribution | Prior to the initial dose on day 1 and 2, 4, 6, 8, 10, 24, and 48 hours post-dose
Time to Disease Progression | end of study
Recommended phase II dose (RP2D) and the optimal dose schedule | End of study
Measurement of intratumoral and skin concentration of sunitinib | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henk MW Verheul, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Rovithi M, Gerritse SL, Honeywell RJ, Ten Tije AJ, Ruijter R, Peters GJ, Voortman J, Labots M, Verheul HMW. Phase I Dose-Escalation Study of Once Weekly or Once Every Two Weeks Administration of High-Dose Sunitinib in Patients With Refractory Solid Tumors. J Clin Oncol. 2019 Feb 10;37(5):411-418. doi: 10.1200/JCO.18.00725. Epub 2018 Dec 26. PMID 30586316